CLINICAL TRIAL: NCT01122186
Title: Intervention Targeting Medication Adherence and Methamphetamine Use in HIV Positive Men
Brief Title: Intervention Targeting Medication Adherence and Methamphetamine Use in HIV Positive Men (ACE)
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Jeffrey T. Parsons, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA023395 (NIH)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: HIV Medication Adherence; Methamphetamine Use; Sexual Risk; Poly-substance Use; HIV Infections
Keywords: Medication Adherence; Methamphetamine Use; Sexual Risk; Poly-substance Use; HIV; Treatment; Motivational Interviewing; Cognitive Behavioral Skills Training; Men Who Have Sex With Men
MeSH Terms: conditions — HIV Infections; Medication Adherence; Homosexuality | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Condition (Experimental): Eight sessions of Motivational Interviewing and Cognitive Behavioral Skills Training, adapted to target both MA use and medication adherence, as well as sexual risk behaviors and polydrug use.
  Interventions: Behavioral: Motivational Interviewing + Cognitive Behavioral Skills Training
- Education Condition (Active Comparator): Eight sessions of education with content designed to mirror the information covered in the intervention condition. The content will be as follows: 3 sessions focusing on medication adherence; 3 sessions focusing on the dangers of methamphetamine use; 1 session addressing sexual risk; and 1 session addressing poly-substance use.
  Interventions: Behavioral: Education Attention Control

INTERVENTIONS:
Behavioral: Motivational Interviewing + Cognitive Behavioral Skills Training — The first two sessions will be primarily Motivational Interviewing and begin with an introduction to the nature of treatment, emphasizing the client's autonomy, and explain that the purpose of the sessions is to explore feelings about their medication adherence, meth use, and any other issues, with the eventual goal of working towards any changes the client may wish to make. During the third session, the client will complete an individualized functional analysis of recent occasions when the client missed medication, used MA and/or other substances, and engaged in risky sex (not necessarily all at the same time). Sessions four through seven will focus on Cognitive Behavioral Skills Training for adherence, reducing or stopping meth use, reducing or stopping the combination of meth and other drug use, and avoiding risky sexual behavior. The final session emphasizes maintenance of behavior change and relapse prevention.
  Arms: Intervention Condition
Behavioral: Education Attention Control — During the first two sessions participants watch the documentary "Rock bottom" to receive information on Crystal Methamphetamine, and the possible interactions between HIV medications and recreational substances. Sessions 3 and 4 focus on the importance of medication adherence, viral replication and mutation, and resistance. Session 5 focuses on the negative effects of several recreational substances as well as the negative effects of mixing substances. Session six discusses HIV stigma, transmission risk sexual behavior, and HIV disclosure. Session 7 revisits medication adherence, focusing on dealing with medication side effects and communicating with health care providers. The final session uses part of the documentary "Meth" which highlights issues of methamphetamine use through interviews with men in various stages of recovery.
  Arms: Education Condition

SUMMARY:
The primary aim is to test an innovative 8-session intervention, based on Motivational Interviewing and Cognitive Behavioral Skills-Training for the co-occurrence of methamphetamine use and highly active antiretroviral therapy (HAART) non-adherence among methamphetamine using HIV+ MSM in NYC, compared to an 8-session educational (ED) condition. Participants in the intervention condition will report greater reductions in the number of days of methamphetamine use and viral load, and greater increases in CD4 counts and self-reported and objectively measured adherence than those in the education condition.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ (confirmed at baseline through documentation)
* Biologically male
* report sex with another man at least once
* report methamphetamine use at least three times in the past three months
* report less than 90% HAART medication adherence, as measured by the total number of days a participant missed an HIV medication in the last 30
* able to communicate with staff and complete a survey that is in English.

Exclusion Criteria:

* Unstable, serious psychiatric symptoms
* Currently suicidal/homicidal
* Evidence of gross cognitive impairment
* Self-reported current enrollment in a drug or HIV-related intervention or research study.
* Methadone use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Adherence to HIV medication | every three months over the course of a year
  Participants in the intervention condition will report greater reductions in viral load, and greater increases in CD4 counts and self-reported adherence than those in the education comparison at at the end of the intervention period (3 months). Those in the intervention condition will also maintain greater reductions in viral load, and greater increases in CD4 counts and self-reported adherence than those in the education comparison condition at the three follow-up assessments (6, 9, and 12 months).
Methamphetamine use. | every three months over the course of a year
  Participants in the intervention condition will report greater reductions in self-reported days of methamphetamine use than those in the education comparison at at the end of the intervention period (3 months). Those in the intervention condition will also maintain greater reductions in self-reported days of methamphetamine use than those in the education comparison condition at the three follow-up assessments (6, 9, and 12 months).

SECONDARY OUTCOMES:
Sexual Risk | every three months over the course of a year
  Participants in the intervention condition will report greater reductions in high-risk sexual behavior compared to participants in the educational comparison condition.
Polysubstance use | every three months over the course of a year
  Participants in the intervention condition will report greater reductions in the use of substances other than methamphetamine, compared to participants in the educational comparison condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for HIV/AIDS Educational Studies and Training of Hunter College, CUNY, New York, New York, United States

REFERENCES:
- See also: Center for HIV/AIDS Educational Studies and Training website — http://www.hunter.cuny.edu/chest/